CLINICAL TRIAL: NCT02336919
Title: The Use of Text Messaging to Improve the Hospital-community Transition and Prevent Readmission in Patients With Cardiovascular Disease (Txt2Prevent)
Brief Title: The Use of Texting Messaging to Improve the Hospital-to-community Transition Period in Cardiovascular Disease Patients
Acronym: Txt2Prevent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Providence Health & Services (Other); University of British Columbia (Other); McMaster University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Scott Lear, Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H14-02385
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Disease; Acute Coronary Syndrome
Keywords: discharge; mHealth; telehealth; text messaging
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Txt2Prevent (Experimental): The treatment group will receive all the usual discharge treatment, instructions and information for acute coronary syndrome patients as well as the Txt2Prevent text-messaging program. The program will include a variety of topics such as standard follow-up care reminders as well as general self-management and healthy living texts. There will be two streams, one for current/recent smokers and one for non-smokers. Texts will be sent out every 1-3 days for 60 days. All participants in the same stream will receive the same texts in the same order.
  Interventions: Behavioral: Txt2Prevent
- Usual Care (No Intervention): The usual care group will receive all standard discharge treatment, instructions and information for patients with acute coronary syndrome, but no text-messaging program. Nurses typically go over important information with patients before they leave as well as give them printed materials.

INTERVENTIONS:
Behavioral: Txt2Prevent — A 60-day text messaging program called Txt2Prevent (see description in the arm description).
  Arms: Txt2Prevent

SUMMARY:
Participants will be recruited during their hospitalization for either heart attack or unstable angina and will be randomly assigned to either a text message program (Txt2Prevent) or usual care. They will be texted for the first 60-days after discharge. Texts will include topics regarding self-management and discharge protocols such as reminders to make an appointment with their general practitioner or to refill medication prescriptions. After 60 days, the two groups will be compared for hospital readmission rates, quality of life, medication adherence, and self-management.

DETAILED DESCRIPTION:
Cardiovascular disease is one of the leading causes for hospitalization and death in Canada. Being discharged is often a challenging and overwhelming time. Sometimes patients are readmitted to the hospital shortly in the months following their discharge. Some of these readmissions are due to information transfer being poor or insufficient.

Previous studies have looked at whether text messaging can be a simple, cost-effective way to help patients. Therefore, we wish to investigate the effectiveness of using text messaging to help heart patients after they are discharged from the hospital.

The goal of this study is to determine the impact of a pilot text-messaging intervention program (Txt2Prevent) that supports coronary syndrome (heart attack and unstable angina) patients for 60 days after their hospital discharge. The program will include information about follow-up care, medication use, and healthy lifestyle behaviours. The texts will be sent at relevant times during the patients' recovery.

The primary objective is compare self-management between the usual care patients versus the Txt2prevent patients. We hypothesize that the Txt2Prevent group will have better self-management than the usual care group.

The secondary objective is compare medication adherence, and health-related quality of life as well as readmission and mortality rates between the two patient groups. We hypothesize that the Txt2Prevent group will have better outcomes for these variables.

The study population is acute coronary syndrome patients at St. Paul's hospital who are discharged. Participants will be randomly assigned to one of two groups-a usual care group and the usual care plus the Txt2Prevent text messaging program group. All participants will undergo a baseline assessment that includes:

* Demographics, medical history, medication use and technology use information
* Self-management skills
* Health-related quality of life

After 60 days, participants will be contacted again to perform a follow up assessment that includes:

* Information on readmission, medication use, the use of health services such as cardiac rehab
* Self-management skills
* Health-related quality of life
* Medication adherence

In both the baseline and follow-up assessments, information may be obtained from the patient's medical chart or records (e.g. medical history) or self-report.

After the intervention, some intervention participants will be contacted to complete a semi-structured interview about their experiences with the Txt2Prevent program.

ELIGIBILITY:
Inclusion Criteria:

* are an acute coronary syndrome patient on the non-surgical ward who will be discharged home
* own a phone with text-messaging capabilities and have the ability to access new text messages
* have the ability to provide informed consent
* have the ability to read and understand English

Exclusion Criteria:

* have a pre-scheduled surgical procedure within the duration of the study
* if it is expected that they will not survive the duration of the study due to non-cardiovascular reasons
* are currently enrolled in another research project regarding CVDs that would interfere with the study outcomes.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Self-management as measured by the Health Education Impact Questionnaire by Osborne et al. | Pre- and post-study period (0 and 60 days)

SECONDARY OUTCOMES:
Medication Adherence as measured by the Morisky Medication Adherence Scale by Morisky et al. | Post-study period (60 days)
Health-related quality of life as measured by the EuroQoL 5D-5L by the EuroQoL group | Pre- and post-study period (0 and 60 days)
Hospital readmissions | Assessed at the end of the study (day 60)
Mortality | Assessed at the end of the study (day 60)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lear, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ross ES, Sakakibara BM, Mackay MH, Whitehurst DGT, Singer J, Toma M, Corbett KK, Van Spall HGC, Rutherford K, Gheorghiu B, Code J, Lear SA. The Use of SMS Text Messaging to Improve the Hospital-to-Community Transition in Patients With Acute Coronary Syndrome (Txt2Prevent): Results From a Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 May 14;9(5):e24530. doi: 10.2196/24530. PMID 33988519
- [Derived] Ross ES, Sakakibara BM, Mackay MH, Whitehurst DG, Singer J, Toma M, Corbett KK, Van Spall HG, Rutherford K, Gheorghiu B, Code J, Lear SA. The Use of Text Messaging to Improve the Hospital-to-Community Transition in Acute Coronary Syndrome Patients (Txt2Prevent): Intervention Development and Pilot Randomized Controlled Trial Protocol. JMIR Res Protoc. 2017 May 23;6(5):e91. doi: 10.2196/resprot.6968. PMID 28536088